CLINICAL TRIAL: NCT01731756
Title: Effects of Leaf Extract of Azadirachta Indica in Palmer Arsenical Keratosis: Randomized, Double Blind, Placebo-controlled Trial
Brief Title: Effects of Leaf Extract of Azadirachta Indica in Palmer Arsenical Keratosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Prof. Mir Misbahuddin, Prof. and Chairman, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BSMMU-003-CT
Record Dates: First submitted 2012-11-16; First posted 2012-11-22 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Arsenical Keratosis
Keywords: Palm; Arsenic; Keratosis; Salicylic acid; Azadirachta indica; Neem
MeSH Terms: conditions — Keratosis | interventions — Salicylic Acid; Petrolatum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palmer arsenical keratosis (study) (Experimental): Leaf extract of A. indica plus salicylic acid (6%) in petroleum jelly base will be applied on palmer keratotic lesion once daily at bedtime for 12 weeks
  Interventions: Other: Leaf extract of A. indica; Drug: Salicylic Acid (6%); Other: Petroleum jelly
- Palmer arsenical keratosis (control) (Placebo Comparator): Salicylic acid (6%) in petroleum jelly base will be applied on palmer keratotic lesion once daily at bedtime for 12 weeks
  Interventions: Drug: Salicylic Acid (6%); Other: Petroleum jelly

INTERVENTIONS:
Other: Leaf extract of A. indica — Leaf extract of A. indica plus 6% salicylic acid will be applied on palmer keratotic lesion once daily at bedtime for 12 weeks.
  Arms: Palmer arsenical keratosis (study)
Drug: Salicylic Acid (6%) — Salicylic acid (6%) will be applied on palmer keratotic lesion once daily on bedtime for 12 weeks.
Other: Petroleum jelly — Petroleum jelly will be applied on palmer keratotic lesion once daily at bedtime for 12 weeks.

SUMMARY:
Effects of leaf extract of Azadirachta indica in palmer arsenical keratosis: Randomized, double-blind, placebo-control trial

DETAILED DESCRIPTION:
The objective of this study is to evaluate the effectiveness of topical administration of the Leaf of Azadirachta indica in the treatment of palmer arsenical keratosis. Fifty patients of moderate palmer arsenical keratosis patients from an arsenic affected area will be recruited on the basis of inclusion and exclusion criteria and had been drinking arsenic contaminated water for more than six months. They will be divided into two groups each will consist of twenty five members. One group will be provided A. indica plus 6% salicylic acid ointment to apply on palm overnight daily for 12 weeks. Another group will be provided 6% salicylic acid ointment . Water and nail sample will be collected before starting recruitment to confirm diagnosis. Then again nail sample will be collected before and after the study to see the level of arsenic in skin. Effects will be observed after every two weeks and change will be detected as nil, mild reduction, moderate reduction and fully cured.

ELIGIBILITY:
Inclusion Criteria:

* Palmer arsenical keratosis
* Drinking arsenic contaminated water (>50 ppb) for more than six months
* Patient voluntarily agree to participate

Exclusion Criteria:

* Pregnancy
* Lactating mother
* Diabetes mellitus
* Rheumatoid arthritis
* Systemic lupus erythematosus
* Psoriasis
* Bowen's disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Changes in palmer arsenical keratosis | 0 week (baseline), 12 weeks (end)
  Size and number of keratotic lesions will be reduced. These will be expressed in score.

SECONDARY OUTCOMES:
Changes in arsenic level in nail | 0 week (baseline), 12 weeks (end)
  Arsenic level in nail of the patient will be decrease. Total arsenic level will be estimated by atomic fluorescence spectrometer.

CONTACTS AND LOCATIONS:
Overall Officials: Mir Misbahuddin, MBBS, PhD, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Department of Pharmacology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh